CLINICAL TRIAL: NCT01574482
Title: Effects of the Consumption of a Plant Sterols-enriched Dairy Fermented Product on Hypercholesterolemia Management in Hypercholesterolemic Adults
Brief Title: Effect of the Consumption of a Fermented Milk Enriched With Plant Sterols (Italy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU216
Record Dates: First submitted 2012-04-07; First posted 2012-04-10 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Mildly Hypercholesterolemic Subjects
Keywords: Plant sterol - Hypercholesterolemia - diet - dairy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Experimental)
  Interventions: Other: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols).
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters

INTERVENTIONS:
Other: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols). — 1 = Intervention 1 (1 test product/day)
  Arms: 1 = Tested product
Other: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters — 2 = Intervention 2 (1 control product/day)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to investigate the cholesterol lowering effect of a drinkable low fat fermented milk enriched with plant sterol after 3 and 6 weeks of daily consumption in mildly hypercholesterolemic people treated or not by statins

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 20-75 years; BMI between 19 and 30 kg/m2 , LDL-cholesterol plasma level between 130 mg/dL to 190 mg/dL (bounds included) with or without any statin monotherapy, with stabilized hypercholesterolemia (since more than 3 months), accepting to follow the dietary recommendations advisable for hypercholesterolemic patient (NCEP-ATP III guidelines), used to consume dairy products, agreeing to a written informed consent, for female: effective contraceptive methods used

Exclusion Criteria:

* Subject with plasma triglycerides (TG) levels > or = 350 mg/dL, with any cardiovascular event in the last 6 months, Subject taking any drugs affecting lipid metabolism (including hypocholesterolemic treatment) other than statin in monotherapy, Diabetic (type I and type II), smoking strictly more than 20 cigarettes/day, presenting known allergy or hypersensitivity to milk proteins, and soy, receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters, with renal failure or any other metabolic disorder which could interfere with the evaluation of efficiency or safety of the product , pregnant and breast feeding women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Silvestrini, Perugia, Italy